CLINICAL TRIAL: NCT06309251
Title: Clinical and Nutritional Effectiveness and Impact on the Quality of Life of the Ketogenic Diet in Pediatric Patients With Neurological, Genetic or Metabolic Disorders: a Multicenter Prospective Observational Study
Brief Title: Effectiveness and Impact on the Quality of Life of Ketogenic Diet in Pediatric Patients
Status: Recruiting | Type: Observational
Sponsor: Danone Nutricia SpA Società Benefit (Industry)
Responsible Party: Sponsor
Other Study IDs: KetoSTrENgTH
Record Dates: First submitted 2024-02-29; First posted 2024-03-13 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Drug Resistant Epilepsy; Autism Spectrum Disorder; Chronic Migraine; Brain Tumor, Pediatric
MeSH Terms: conditions — Drug Resistant Epilepsy; Autism Spectrum Disorder; Brain Neoplasms | interventions — Diet, Ketogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients requiring KD: Pediatric patients with any disease which require a ketogenic diet (KD), i.e. metabolic or genetic disorder or neurological (congenital and acquired) diseases
  Interventions: Other: ketogenic diet (as per clinical practice)

INTERVENTIONS:
Other: ketogenic diet (as per clinical practice) — Patients recruited receive a ketogenic diet. The prescription, the type of KD protocol and the route of administration will depend, essentially, on the patient's ability and willingness to feed spontaneously and independently, as well as on compliance with the therapies set and the severity of the clinical conditions.

SUMMARY:
The goal of this observational study is to learn about the clinical and nutritional effectiveness of ketogenic diet (KD) in pediatric patients with genetic, neurological or metabolic conditions requiring KD.

The main question[s] it aims to answer are:

* does KD support adequate growth?
* does KD improve clinical symptoms?
* how does KD impact quality of life? Participants will be followed up as per clinical practice

DETAILED DESCRIPTION:
Scientific and clinical interest in KD is growing with a progressive increase in its therapeutic indications, ie recent studies show beneficial effects of KD in other diseases like migraine, autism spectrum disorder and brain tumors.

However, so far, the majority of results on KD effects have been collected in patients with drug-resistant epilepsy proving its effectiveness on clinical outcome (e.g. reducing epileptic seizures), frequently leaving out the nutritional assessment and the impact on quality of life. Nonetheless, these factors are indeed essential to ensure safety and efficacy of KD treatment, especially when dealing with children and in perspective of the progressive expansion of the target population that can benefit from this nutritional therapy.

The present multicenter study aims to analyse these poorly explored areas, by evaluating, in a cohort of pediatrics patient with indication to KD therapy, not only the KD effectiveness on the course of the underlying disease, but also the impact on nutritional parameters (e.g. growth, lipid profile, vitamin intake, bone mineral density, ..) and on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (aged < 18 years) with drug-resistant epilepsy (fail to achieve (and maintain) seizure freedom with adequate trials of two or more antiseizure medications) or genetic, metabolic, neurological (congenital and acquired) diseases treated with ketogenic diet
* Pediatric patients (aged < 18 years) with metabolic, genetic or neurological (congenital and acquired) diseases (not necessarily associated with drug-resistant epilepsy) treated with ketogenic diet; this includes the new KD indications or the administration of KD in the ICU for status epilepticus.

Exclusion Criteria:

* Patients affected by beta-oxidation cycle disorders, systemic primary carnitine deficiency, primary dyslipidemia, pyruvate carboxylase deficiency, porphyria, mitochondrial disease, defects in ketone body metabolism (ketogenesis or ketolysis), defect in gluconeogenesis.
* Children with type 1 diabetes
* Parents (or caregivers) unable to guarantee adherence to the

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatri patients (0-18 years) affected by any disease which require a ketogenic diet (KD), i.e. metabolic or genetic disorder or neurological (congenital and acquired) diseases
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Nutritional adequacy | 6 months
  evaluate the nutritional adequacy of the diet after 6 months of treatment with ketogenic diet (KD) in terms of adequate growth defined by weight-for-age Z Score (WAZ) and length-for-age Z score (LAZ).

SECONDARY OUTCOMES:
Nutritional adequacy | 6 months,(12 months optional)
  Evaluate the nutritional adequacy of the diet after 6 and 12 months of treatment with ketogenic diet (KD) in terms of correct growth defined by:
  Weight-for-age Z-score (WAZ), length/height-for-age z-score (LAZ), BMI z-score Blood levels of selected parametres (eg cholesterol, HDL, LDL) within normal ranges Body composition (optional)
% of responders to KD | 6 months,(12 months optional)
  Evaluate the effectiveness of the ketogenic diet (KD) on the clinical outcomes (% of responders):
  * Epilepsy: at least 50% seizure reduction after 6 months of KD treatment (vs 6 months before trial start( (daily diary records)
  * ASD: reduction of at least 2-8 in CARS score after 6 months of KD treatment
  * Chronic migraine: at least 50% episodes reduction after 6 months of KD treatment (vs 6 months before trial start( (daily diary records); reduction >=50% of PedMiDas score after 6 months of KD treatment (vs baseline) Brain tumors: % survival; % of subjects with progression free survival
Health related quality of life improvement through parent questionnaire | 6 months,(12 months optional)
  Evaluate the effectiveness of the ketogenic diet (KD) on the patient's quality of life using a non-validated questionnaire administered to parents with qualitative open and closed questions. Improvement will be considered as an improvement in the score of disease burden related questions baseline vs end of observation

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - ASST Fatebenefratelli Sacco (PO "V. Buzzi"), Milan, MI
  - Fondazione "Istituto Neurologico Nazionale C. Mondino", Pavia, PV
  - Ospedale Pediatrico Bambino Gesù, Roma, RM

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bertoli S, Foppiani A, De Amicis R, Leone A, Mastella C, Bassano M, Giaquinto E, Baranello G, Battezzati A. Anthropometric measurement standardization for a multicenter nutrition survey in children with spinal muscular atrophy. Eur J Clin Nutr. 2019 Dec;73(12):1646-1648. doi: 10.1038/s41430-019-0392-2. Epub 2019 Jan 15. PMID 30647441
- [Background] Cole TJ, Flegal KM, Nicholls D, Jackson AA. Body mass index cut offs to define thinness in children and adolescents: international survey. BMJ. 2007 Jul 28;335(7612):194. doi: 10.1136/bmj.39238.399444.55. Epub 2007 Jun 25. PMID 17591624
- [Background] Hershey AD, Powers SW, Vockell AL, LeCates S, Kabbouche MA, Maynard MK. PedMIDAS: development of a questionnaire to assess disability of migraines in children. Neurology. 2001 Dec 11;57(11):2034-9. doi: 10.1212/wnl.57.11.2034. PMID 11739822
- [Background] Kossoff EH, Zupec-Kania BA, Auvin S, Ballaban-Gil KR, Christina Bergqvist AG, Blackford R, Buchhalter JR, Caraballo RH, Cross JH, Dahlin MG, Donner EJ, Guzel O, Jehle RS, Klepper J, Kang HC, Lambrechts DA, Liu YMC, Nathan JK, Nordli DR Jr, Pfeifer HH, Rho JM, Scheffer IE, Sharma S, Stafstrom CE, Thiele EA, Turner Z, Vaccarezza MM, van der Louw EJTM, Veggiotti P, Wheless JW, Wirrell EC; Charlie Foundation; Matthew's Friends; Practice Committee of the Child Neurology Society. Optimal clinical management of children receiving dietary therapies for epilepsy: Updated recommendations of the International Ketogenic Diet Study Group. Epilepsia Open. 2018 May 21;3(2):175-192. doi: 10.1002/epi4.12225. eCollection 2018 Jun. PMID 29881797